CLINICAL TRIAL: NCT04908371
Title: Selective Trunk Block Versus Hybrid Interscalene-Supraclavicular Brachial Plexus Block for Anaesthesia of the Entire Upper Extremity: A Randomized Double-Blind Controlled Trial
Brief Title: Selective Trunk Block vs Hybrid Interscalene Supraclavicular BPB for Anaesthesia of the Entire Upper Extremity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Published data indicated Selective Trunk Block is a better choice
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SeTB vs IS-SC Ver2
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Selective Trunk Block; Hybrid Interscalene-Supraclavicular Brachial Plexus Block
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Pharmaceutical Preparations; Lidocaine; Epinephrine; Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive either a SeTB (SeTB group) or hybrid interscalene-supraclavicular BPB (IS-SC group) under ultrasound guidance. The randomization sequence will be generated using an online randomization software (www.randomization.com). The randomization sequence will be assigned as 1 = selective trunk block (SeTB group) and 2 = interscalene-supraclavicular BPB (IS-SC group). The group allocation will be prepared by a computer officer (third party) in the Department of Anaesthesia & Intensive Care, of the Chinese University of Hong Kong.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients in both study groups will not be able to see the ultrasound monitor during block placement and therefore will be blinded to group allocation. The "outcome assessor" (research nurse) will not be present in the procedure room during block placement and thus will also be blinded to group allocation. Dressings applied on the skin to cover the needle entry sites will also be identical in the two study groups. The anaesthesiologist (principal investigator) performing the allocated BPB will take no further part in the study after block placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Trunk Block (SeTB) (Active Comparator): Patients will lie flat on their back on the examination couch with the arm in neutral position and the head turned slightly to the opposite side. Ultrasound scan will be performed sequentially starting from the base of the neck (supraclavicular fossa) to the upper part of the interscalene groove and then in the reverse direction to the supraclavicular fossa. After identifying the three trunks of the brachial plexus, ultrasound guided selective trunk block will be done using local anesthetic agents (a mixture of 2% lidocaine with 1:200,000 epinephrine and 0.5% levobupivacaine in a total of 20ml) will be injected at the superior, middle, and inferior trunks of the brachial plexus in order to anesthetize the whole upper limb.
  Interventions: Procedure: Selective Trunk Block
- Interscalene-Supraclavicular Brachial Plexus Block (IS-SC-BPB) (Active Comparator): Patients will lie flat on their back on the examination couch with the arm in neutral position and the head turned slightly to the opposite side. Ultrasound scan will be performed sequentially starting from the base of the neck (supraclavicular fossa) to the upper part of the interscalene groove. The unique sonomorphology of the C7 transverse process will be used as the key anatomical landmark to identify the individual elements of the brachial plexus. Under ultrasound guidance, local anesthetic agents (a mixture of 2% lidocaine with 1:200,000 epinephrine and 0.5% levobupivacaine in a total of 30ml) will be injected at the interscalene groove and at the supraclavicular fossa in order to anesthetize the whole upper limb.
  Interventions: Procedure: Interscalene-Supraclavicular Brachial Plexus Block (IS-SC BPB)

INTERVENTIONS:
Procedure: Selective Trunk Block — It is one type of peripheral nerve blocks for upper extremity surgery. Patients will have an ultrasound scan and nerve block with local anesthetic (LA) agent (a mixture of 2% Xylocaine with 1:200,000 adrenaline and 0.5% Chirocaine in a total of 20ml) injected at the trunks of the brachial plexus in order to produce the anesthesia of the whole upper extremity of the patients scheduled for upper limb surgery. SeTB will be performed as a "two-injection technique". One at the side of the neck (interscalene groove) of the affected upper limb, injections will be made near the superior trunk (5mL) and follow by redirection of the needle under ultrasound guidance to inject the LA to middle trunk (5mL). Then the second skin puncture will be made near the upper part mid-collar bone (supraclavicular fossa) to inject the LA to the inferior trunk (10mL).
  Other Names: Drug (Xylocaine with adrenaline and Chirocaine)
  Arms: Selective Trunk Block (SeTB)
Procedure: Interscalene-Supraclavicular Brachial Plexus Block (IS-SC BPB) — It is another type of peripheral nerve blocks for upper extremity surgery. Patients will have an ultrasound scan and nerve block with local anesthetic (LA) agent (a mixture of 2% Xylocaine with 1:200,000 adrenaline and 0.5% Chirocaine in a total of 30ml) injected at the interscalene groove and supraclavicular fossa, so "two-injection technique" will be adopted. The first skin puncture will be near the side of the neck (interscalene groove) of the affected upper limb (15mL) and then the second skin puncture will also be made near the upper mid-collar bone (supraclavicular fossa) to inject 15mL of LA.
  Other Names: Drug (Xylocaine with adrenaline and Chirocaine)
  Arms: Interscalene-Supraclavicular Brachial Plexus Block (IS-SC-BPB)

SUMMARY:
The objective of this study is to compare the clinical effectiveness in producing anesthesia of the whole upper limb between two regional blocks - Selective Trunk Block (SeTB) and Hybrid Interscalene Supraclavicular Brachial Plexus Block (hybrid IS-SC BPB).

DETAILED DESCRIPTION:
Brachial plexus block (BPB) is frequently used as the sole anesthestic technique for upper extremity surgery. The choice of injection can be made from different approaches that often depends on the site of surgery because the extent of sensory-motor blockade after a BPB varies with the approach used. However, there is no single BPB technique that can consistently produce anesthesia of the whole ipsilateral upper extremity. Nevertheless, cases such as combined fracture of the upper humerus and forearm bones have to anesthetize the whole upper extremity for surgery or those with multiple comorbidities and unfit for general anesthesia. In these cases, multiple injections have to be made. Thus, a combined ultrasound guided (USG) interscalene-supraclavicular (IS-SC) BPB has to be used as the sole anesthetic for proximal humerus surgery but with a relatively large volume (35-50mL) of numbing medication, which often exceed the recommended maximum safety dose. Recently principal investigator has demonstrated that it is feasible to accurately identify majority of the main components of the brachial plexus above the clavicle, including the three trunks, using ultrasound imaging. As majority of the innervation of the upper extremity, i.e. shoulder, arm, elbow, forearm, wrist and hand, originates from the three trunks of the brachial plexus, principal investigator has proposed that selectively blocking the superior, middle and inferior trunks of the brachial plexus under ultrasound guidance, will produce anesthesia of the entire upper limb. Principal investigator refers this technique as selective trunk block (SeTB). The preliminary experience with SeTB for anesthesia of the entire upper limb with smaller volumes (25ml) of numbing medication is feasible and able to ensure total immobility of the whole upper limb that meets the essential requirement for surgery. In this study principal investigator hypothesizes that USG guided SeTB is not inferior to USG IS-SC BPB in terms of its ability to produce sensory-motor blockade.

The aim of this study is to compare the proportion of patients who develop "readiness for surgery" for 30 minutes between a SeTB and hybrid IS-SC BPB. In other words, comparing the clinical effectiveness in producing anesthesia of the whole ipsilateral upper limb between SeTB and hybrid IS-SC brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I-III
* undergoing elective or emergency upper extremity surgery involving the proximal humerus to distal hand or surgery involving any combination of these regions scheduled for a brachial plexus block

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Skin infection at the site of block
* History of allergy to local anesthetic agents
* Bleeding tendency or with evidence of coagulopathy
* Pre-existing neurological deficit or neuromuscular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Readiness for surgery | within 45 minutes after the block at 5 minutes interval
  An overall sensory score of =<30 (loss of sensation to cold stimulus (ice cube), NRS: 100-0, 100=normal sensation, 0=no sensation) and motor score of =<1 (3-points scale: 2=no block, 1=paresis, 0=paralysis) in all the nerves (C5 to T1) tested.
  Sensation block assessment: C5 - lateral (radial) side of the antecubital fossa (just proximal to elbow crease), C6 - thumb, dorsal surface, proximal phalanx, C7 - middle finger, dorsal surface, proximal phalanx, C8 - little finger, dorsal surface, proximal phalanx, and T1 - medial (ulnar side of the antecubital) fossa, just proximal to the medial epicondyle of the humerus.
  Motor block assessment: C5 - elbow flexors (biceps, brachialis), C6 - wrist extensors (extensor carpi radialis longus and brevis), C7 - elbow extensors (triceps), C8 - finger flexors (flexor digitorum profundus) to the middle finger, T1 - small finger abductors (abductor digiti minimi).
Complete sensory-motor block | within 45 minutes after the block at 5 minutes interval
  An overall sensory score and motor score of '0'. Sensation to coldness (ice) with sensory score of '0' [sensory score 100-0: sensory 100=normal sensation, and 0=no sensation] for C5 - lateral (radial) side of the antecubital fossa (just proximal to elbow crease), C6 - thumb, dorsal surface, proximal phalanx, C7 - middle finger, dorsal surface, proximal phalanx, C8 - little finger, dorsal surface, proximal phalanx, and T1 - medial (ulnar side of the antecubital) fossa, just proximal to the medial epicondyle of the humerus.
  Motor blockade will be graded using a 3-point scale: 2=no change, 1=reduced contraction (paresis), 0=paralysis. Motor block assessment at C5 - elbow flexors (biceps, brachialis), C6 - wrist extensors (extensor carpi radialis longus and brevis), C7 - elbow extensors (triceps), C8 - finger flexors (flexor digitorum profundus) to the middle finger, T1 - small finger abductors (abductor digiti minimi).

SECONDARY OUTCOMES:
Changes of sensory block of each nerve (C5 to T1) | within 45 minutes after the block at 5 minutes interval
  The time it takes to achieve a sensory block score of =<30 (loss of sensation to cold stimulus (ice cube), NRS: 100-0 100=normal sensation, 0=no sensation).
  C5 - lateral (radial) side of the antecubital fossa (just proximal to elbow crease), C6 - thumb, dorsal surface, proximal phalanx, C7 - middle finger, dorsal surface, proximal phalanx, C8 - little finger, dorsal surface, proximal phalanx, and T1 - medial (ulnar side of the antecubital) fossa, just proximal to the medial epicondyle of the humerus.
Changes of motor block of each nerve (C5 to T1) | within 45 minutes after the block at 5 minutes interval
  The time it takes to achieve a motor block score of =<1 (3-point motor grade: 2=no change, 1=reduced contraction (paresis), 0=paralysis).
  C5 - elbow flexors (biceps, brachialis), C6 - wrist extensors (extensor carpi radialis longus and brevis), C7 - elbow extensors (triceps), C8 - finger flexors (flexor digitorum profundus) to the middle finger, T1 - small finger abductors (abductor digiti minimi).
Block performance time | within 30 minutes after entering the procedure room
  the time taken from the start of the local anesthetic (LA) skin infiltration to the end of the LA injection for the block
Discomfort score | immediately after the end of the block
  Discomfort experienced during the regional anesthesia using a numeric rating scale (NRS, 0 to 100, 0=no discomfort, 100=extreme discomfort)
Paresthesia | immediately after the end of the block
  Any paresthesia experienced during the block will be assessed and recorded as a 'yes' or 'no' response
Complications | within 45 minutes after the block
  Any complications directly related to brachial plexus block (vascular or pleural puncture, ipsilateral Horner's syndrome, intraneural injection with nerve swelling or symptoms suggestive of local anesthetic toxicity) will be record.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, New Territories, Hong Kong